CLINICAL TRIAL: NCT03900221
Title: French Registry for Monitoring Pregnancies and Children of Women With Multiple Sclerosis Within The Observatoire Français de la Sclérose en Plaque (OFSEP) Cohort
Brief Title: French Registry for Monitoring Pregnancies for Multiple Sclerosis
Acronym: RESPONSE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0631; 2018-A02552-53 (Other: ID-RCB)
Record Dates: First submitted 2019-03-08; First posted 2019-04-02 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Sclerosis, Multiple; Neuromyelitis Optica Spectrum Disorder; Myelin Oligodendrocyte Glycoprotein (MOG)-Antibody Related Disorders; Pregnancy Abnormal
Keywords: Multiple sclerosis; pregnancy; disease modifying drugs; breastfeeding; loco-regional analgesia
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women with multiple sclerosis or related neurological: Children born to women with multiple sclerosis or related neurological syndromes.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The influence of pregnancy on the course of multiple sclerosis (MS) has long been a controversial topic. After the publication of the first large prospective study of pregnancy and MS in 1998, counselling of women with MS has radically changed and many patients have been able to fulfill their desire of motherhood. However, there are still some challenges for the neurologist, who has to face old unanswered questions or new issues, regarding the use of disease modifying drugs (DMDs) in this period of life, effects on the short and long term outcome of the mother (in terms of relapses and disability) and the child, role of breast-feeding and locoregional analgesia.

To set up a national prospective pregnancy registry for patients with MS, nested within the Observatoire Français de la Sclérose en Plaque (OFSEP) cohort, owing to a better knowledge of interactions between MS and pregnancy-related issues (pregnancy itself, locoregional analgesia, breastfeeding, impact of using or stopping DMDs on women/children…)

DETAILED DESCRIPTION:
METHODOLOGY Prospective, observational, multicentric and national epidemiological study, within the scope of the OFSEP, including all groups of patients eligible to participate in the Observatoire Français de la Sclérose en Plaque (OFSEP) (definite MS, radiologically isolated syndromes, clinically isolated syndromes, neuromyelitis optica (NMO) and NMO spectrum disorders), with no age limit and an ongoing pregnancy. Women will be followed during pregnancy and in the year after and their children until 6 years of age.

STATISTICAL ANALYSIS To be determined for each specific question. EXPECTED RESULTS Interactions between pregnancy and MS course have been well characterized before the therapeutic era. Neurologists and patients are lacking information to weigh benefits and risks of DMDs used immediately before or during pregnancy, including short and long-term risks to the mother and to the child, but also after delivery. This study should help provide better answers to those questions as well as to still controversial questions about locoregional analgesia and breastfeeding. By following these patients within the Observatoire Français de la Sclérose en Plaque (OFSEP) cohort, the investigator will also have access to a comprehensive description of MS before pregnancy but also in the long term.

ELIGIBILITY:
Inclusion Criteria:

* All groups of patients eligible to participate to the Observatoire Français de la Sclérose en Plaque (OFSEP), including :
* Definite Multiple sclerosis (MS) according to McDonald criteria
* Whatever the clinical course (single attack MS, relapsing-remitting MS, secondary progressive MS, primary progressive MS)
* Radiologically Isolated Syndromes (RIS) (will be validated by the RIS expert group)
* Clinically Isolated Syndromes (CIS)
* Neuromyelitis optica (NMO) and NMO spectrum disorders (will be validated by the "Neuro-optico-myélite aiguë de Devic et des syndromes neurologiques apparentés" (NOMADMUS) expert group)
* No age limit (patients under the age of 18 might be included, provided informed consent is obtained from the parents)
* Ongoing pregnancy: there will be no limit in the gestational age at inclusion. Women can be included at any time before delivery, but the gestational age at inclusion will be recorded and introduced in the analyses whenever pertinent. However, neurologists and patients will be encouraged to start the study as soon as pregnancy is diagnosed.
* Able to give informed consent
* Able to read and/or understand French

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with multiple sclerosis or related neurological syndromes
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2036-08-12 (Estimated); Study Completion 2036-08-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 during pregnancy period | up to 2 years
  Description of the current neurological practice of French neurologists regarding disease modifying drugs and desire of pregnancy and evaluation of its short term impact on the risk of relapses.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 during post-partum period | up to 2 years
  Description of the current neurological practice of French neurologists regarding disease modifying drugs and desire of pregnancy and evaluation of its short term impact on the risk of relapses.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra VUKUSIC, Prof., Principal Investigator — Hospices Civils de Lyon
Locations (48):
- France (47):
  - Chu D'Amiens, Amiens
  - Centre Hospitalier Annecy Genevois, Annecy
  - Centre Hospitalier d'Avignon, Avignon
  - Hopital Jean Minjoz, Besançon
  - Hopital Pellegrin, Bordeaux
  - Hôpital de Brive, Brive-la-Gaillarde
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - Hopital Cote de Nacre, Caen
  - Centre hospitalier Métropole Savoie, Chambéry
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - Hopital Du Bocage, Dijon
  - Ch Epinal, Épinal
  - Hôpital Raymond Poincaré, Garches
  - Centre hospitalier Joséphine Baker Gonesse, Gonesse
  - Chu de Grenoble, Grenoble
  - Centre Hospitalier de Versailles Hôpital Andre Mignot, Le Chesnay
  - Hôpital St Vincent De Paul, Lille
  - Chru de Lille, Lille
  - Hopital Dupuytren, Limoges
  - Cabinet médical Dr Philippe NEUSCHWANDER, Lyon
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Cabinet médical Dr C. CORNUT-CHAUVINC, Lyon
  - Hopital Timone Adultes, Marseille
  - Hopital Gui de Chauliac, Montpellier
  - Cabinet médical Dr L. GUILLOTON, Mornant
  - Hôpital Central, Nancy
  - Hopital Pasteur, Nice
  - Hopital Caremeau, Nîmes
  - Hôpital Paris Saint Joseph, Paris
  - Fondation Rotschild, Paris
  - Hôpital national des Quinze-Vingt., Paris
  - Hopital Pitie Salpetriere, Paris
  - Chi Poissy Saint Germain En Laye, Poissy
  - Chr La Miletrie, Poitiers
  - Hopital Rene Dubos, Pontoise
  - Hopital Pontchaillou, Rennes
  - Hôpital Charles-Nicolle, Rouen
  - Centre Hospitalier de Saint-Denis, Saint-Denis
  - Hopital G. Et R. Laennec, Saint-Herblain
  - Centre Hospitalier Mémorial, Saint-Lô
  - Hopital Nord, Saint-Priest-en-Jarez
  - Hopital Hautepierre, Strasbourg
  - Hôpital Foch, Suresnes
  - Hopital Purpan, Toulouse
  - Chru de Tours Hopital Bretonneau, Tours
  - Médipôle Lyon Villeurbanne, Villeurbanne
- Hopital P. Zobda-Quitman, Fort-de-France, Martinique

REFERENCES:
- See also: Related Info — http://www.ofsep.org